CLINICAL TRIAL: NCT01938924
Title: A Randomised Control Trial to Establish if Use of the gekoTM (Trademark) Post Infra-inguinal Surgical Vein Revascularisation Increases Flow Through the Graft
Brief Title: Surgical Revascularisation and Nerve Stimulation Trial
Acronym: SRANS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12/YH/0480
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention): No intervention
- GekoTM (Active Comparator): geko applied to bypass limb
  Interventions: Device: GekoTM

INTERVENTIONS:
Device: GekoTM — electrical neuromuscular stimulation
  Arms: GekoTM

SUMMARY:
A study to investigate if the gekoTM device improves flow through vascular bypass grafts

DETAILED DESCRIPTION:
The geko™ device, (CE 558928;British Standards Institute notified body 0086), wearable, discrete, self-contained stimulation unit that adheres to the skin (see www.gekodevices.com). The, geko™ produces small electrical impulses that gently activate the common peroneal nerve within the popliteal fossa, behind the knee, in turn activating the venous muscle pumps of the calf and foot. Substantive increases in lower limb blood flow have been demonstrated to improve arterial, venous and microcirculatory blood flow with no reported morbidity.

RATIONALE Early infra-inguinal graft failure, i.e. occurring within 30 days of surgery occurs in approximately 5% of patients16. It is known that the predominant cause of this is thrombosis. The geko™ is an electrical device placed over the common peroneal nerve alongside the knee. The device activates muscle contraction in the peronei using low intensity, low frequency (1Hz) stimulation. The muscle contraction expresses blood from the deep venous system. Application of the stimulation device over the peroneal nerve is suitable for practical purposes. Previous studies have shown that the geko™ substantively increases arterial, venous and microcirculatory blood flow in healthy volunteers. A significant decrease in Tissue Plasminogen Activator antigen has also been demonstrated which indicates increased fibrinolytic activity3. Application of the geko™ device should therefore decrease stasis and increase flow though the graft and as such reduce the risk of thrombosis and as such graft failure.

Study:

Environmental Conditions The examinations will be carried out in a designated temperature controlled clinical room in the Vascular Lab at Hull Royal Infirmary. Participants will be required to abstain from vigorous exercise, nicotine, caffeine and fatty foods prior to their examination. They will be required to wear light garments with their legs exposed.

The geko™ device will be applied to outer/ posterior aspect of the knee whilst the subjects are semi-recumbent, with their knees flexed. The participants will be given 30 minutes in the quiet, environmentally controlled room prior to commencement of measurement to enable equilibration.

Assessments Participants will complete the McGill Pain questionnaire prior to device activation Participants will have the geko™ device applied whilst semi-recumbent with their knees flexed. The intensity will be increased until visible muscle stimulation is evident (concentric isotonic contractions) or until patient tolerance is reached

* Laser Doppler imaging will be used to assess microcirculation flow on the dorsum of both feet at:

  1. Baseline (rest)
  2. 5 minute intervals while the geko™ device is active
  3. 30 minutes following removal of the device Laser Doppler flowmetry is a reproducible, objective, non-invasive measurement which can be used to evaluate real time cutaneous blood flow. The low powered light is conducted via glass fibres to a probe attached to the skin and is scattered by the movement of blood cells inducing a Doppler shift. This allows information on flux and cell velocity to be recorded. The system to be used for this trial is the Moor Instruments DT-4 mains unit with integrated bilateral lasers.
* Ultrasound Doppler arterial flow velocity and blood volume flow within the femoral artery (mid thigh) bilaterally at:

  1. Baseline (rest)
  2. 30 minutes while the device is active
* Ultrasound Doppler flow velocity in femoral vein (mid thigh) bilaterally at:

  1. Baseline (rest)
  2. 40 minutes while the geko is active
* Vicorder measurements of arterial stiffness, pulse wave velocity and stroke volume at:

  1. Baseline (rest)
  2. Immediately following removal/ deactivation of the device
* Vascular Endothelial Growth Factor (VEGF), Tissue Plasminogen Activator antigen (TPA antigen), Full blood count (FBC) and Plasminogen activator inhibitor-1 (PAI-1): 15 mls of blood to be taken from both femoral veins at:

  1. Baseline (rest)
  2. 45 minutes while the geko™ device is active ELISA analysis will be carried out on samples (see appendix). Vascular Endothelial Growth Factor - Therapies which can lead to the development of new, collateral blood vessels, are of particular interest in the field of peripheral arterial disease where narrowing or blockages in existing blood vessels result in tissue ischaemia. Vascular endothelial growth factor (VEGF) is a signal protein produced by cells that stimulates the growth of new blood vessels from pre-existing vessels. Several previous studies have shown that electrical stimulation increases VEGF levels and in turn increases vessel density in muscles.

Tissue plasminogen activator (tPA) is a protein involved in the breakdown of blood clots. As a result it has therapeutic uses in clinical medicine to treat thromboses and emboli. Electrical stimulation has been previously shown to provoke an acute release of tPA into the circulation, although it appears that this response decreases with repeated stimulations. Use of the geko™ device has been shown to result in a significant decrease in Tissue Plasminogen Activator (tPA) antigen which is indicative of increased fibrinolytic activity.

Plasminogen activator inhibitor- 1 (PAI-1) is the primary inhibitor of plasminogen activators and inactivates tissue plasminogen activator (t-PA) and urokinase-type plasminogen activator (u-PA). PAI-1 is an important inhibitor of the fibrinolytic system, and elevated levels could suppress fibrinolysis and result in an increased risk of thrombosis. Increased PAI-1 levels have been shown to be associated with a number of atherosclerotic risk factors, PAI-1 has been shown to act as a prothrombic factor in both arterial and venous thromboembolic disorders.

* Ankle Brachial Pressure Index at baseline and post removal of geko™- utilising both Posterior Tibial Artery and Anterior Tibial Artery
* Maximum calf circumference at baseline and post removal of geko™
* Three blood pressure and heart rate measurements will be taken bilaterally at baseline and @ 30 minutes while the device is active. The mean of the three values will be used for comparison.
* Patient tolerance/ acceptability + Nurse tolerance/ ease of application Questionnaire using Visual Analogue Scores and Verbal Rating Scores to be completed following removal of geko™ device (see appendix)
* The McGill Pain Questionnaire to be completed following device removal

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years,
2. Undergoing infra-inguinal vein bypass graft.
3. Intact cutaneous sensations to nociception in the lower limb, as determined by the investigator.
4. Intact healthy skin at site of application.
5. On effective contraception if sexually active - oral contraceptive pill (> 3 months use), condoms, intrauterine contraceptive device, depot injection.
6. Able to understand the Patient Information Sheet and capable and willing to give informed consent and follow the protocol requirements

Exclusion Criteria:

1. History of haematological disorder or DVT within the preceding 6 months,
2. Pregnant or planning to become pregnant during study duration,
3. Pacemakers or implantable defibrillators,
4. Use of any other neuro-modulation device,
5. Current use of TENS in pelvic region, back or legs,
6. Use of investigational drug/device therapy within past 4 weeks that may interfere with this study,
7. Significant varicose veins or lower limb ulceration.
8. Recent surgery (such as abdominal, gynaecological, hip knee replacement).
9. Recent trauma to lower limbs.
10. Chronic Obesity (BMI Index >34).
11. Any medication judged to be significant by the Principal Investigator.
12. Any significant illness during the four (4) weeks preceding the screening period of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in arterial blood volume flow in the bypass graft measured by ultrasound. | 1 day
  Measured by ultrasound duplex

SECONDARY OUTCOMES:
To assess effect on blood flow in the superficial femoral vein | 1 day
  Measured by ultrasound doppler
To assess effect on microcirculation | 1 day
  Measured using laser Doppler flowmetry
To assess effect on pulse wave velocity, cardiac output and stroke volume | 1 day
  Measured using using the Vicorder device.
To assess effect on levels of VEGF, PAI-1 and tPA antigen. | 1 day
  Blood tests and ELISA
To assess the impact of gekoTM device on pain score utilising the McGill Pain score | 1 day
  Validated pain questionnaire
Patient tolerance/ acceptability | 1 day
  Questionnaire using Visual Analogue Scores and Verbal Rating Scores to be completed following removal of geko™ device
To assess effect on calf circumference | 1 day
  Measurement pre and post device

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Barnes, MRCS, MA, Study Chair — Hull Royal Infirmary
Locations (1):
- Hull Royal Infirmary, Hull, EastRiding of Yorkshire, United Kingdom